CLINICAL TRIAL: NCT04896450
Title: Comparison of the Guided Tissue Regeneration (GTR) Procedure Alone and in Combination With Immediate Orthodontic Tooth Movement (OTM) in the Treatment of Non-containing and Wide Intrabony Periodontal Defects: a Prospective RCT
Brief Title: Comparison of the GTR Procedure Alone and in Combination With Immediate OTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Schupbach Ltd. (Unknown); Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Pal Nagy, Assistant Professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTHO-GTR
Record Dates: First submitted 2021-04-29; First posted 2021-05-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Intrabony Periodontal Defect
Keywords: guided tissue regeneration; orthodontic tooth movement; histology; bone remodeling; deproteinized bovine bone mineral
MeSH Terms: interventions — Guided Tissue Regeneration; Tooth Movement Techniques

STUDY DESIGN:
Intervention Model Description: Patients undergo GTR procedure, after they are randomly allocated either to test (with OTM) or control group (without OTM)
Who Masked: Outcomes Assessor
Masking Description: The histologist is blinded to the study protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Test subjects receive GTR and early initiation of OTM.
  Interventions: Procedure: Guided tissue regeneration (GTR); Device: Orthodontic tooth movement (OTM)
- Control group (Active Comparator): Control subjects receive only GTR.
  Interventions: Procedure: Guided tissue regeneration (GTR)

INTERVENTIONS:
Procedure: Guided tissue regeneration (GTR) — GTR is handled with the utilization of a coronally advanced flap, followed by a thorough debridement of the denudated root surface and the intrabony component. Regenerative materials are resorbable collagen membrane (BioGide, Geistlich Phara AG, Wolhusen, Switzerland) and deproteinized bovine bone mineral (BioOss, Geistlich Phara AG), finally surgery is finished with multilayer suturing technique.
  Other Names: Regenerative surgery of an intrabony periodontal defect
Device: Orthodontic tooth movement (OTM) — An early initialization of the tooth movement with the help of a multibond fixed orthodontic device utilizing low level of continuous orthodontic forces.
  Other Names: Multibond fixed orthodontic appliance
  Arms: Test group

SUMMARY:
The aim is to evaluate in a prospective, randomized, controlled clinical study the healing of a GTR procedure, when it is combined with an immediate orthodontic tooth movement or used alone. Clinical, radiological and reentry (histological) evaluation of a regenerative surgical method (GTR + grafting material) with different postsurgical healing patterns in the treatment of wide, non-containing intrabony defects.

DETAILED DESCRIPTION:
There is limited histological data in literature on the behavior of xenogeneic graft materials in intrabony defects used in periodontal regenerative therapy followed by orthodontic tooth movement (OTM). This clinical study aims to clinically and histologically evaluate the healing response of the periodontal tissues and the healing pattern of a non-resorbable graft material, when they are exposed to orthodontic forces. Therefore teeth presenting non-contained intrabony defects in combination with pathologic tooth migration (PTM) are included in this prospective clinical study. Guided tissue regeneration (GTR) with the application of deproteinized bovine bone mineral (DBBM) and a resorbable collagen membrane is utilized to surgically treat the periodontal defects, which is followed by a random allocation of the patients into test or control group. Subject teeth undergo an early initiated orthodontic treatment after surgery or stay splinted without any tooth movement in the latter groups, respectively. Teeth in test group can be further divided into subgroups, depending if they are moved toward to the former defect (pressure site) or moved away from the defect (tension site). After 9 months of healing a reentry surgery is performed, when a biopsy core is removed with a microtrephine from the previous defect site. The sample is evaluated by means of histology supplemented with histomorphometry, which is the primary outcome variable. Periodontal clinical parameters measured at baseline and at 9 months serves for secondary outcomes. Several studies confirmed the success of graft materials in such comprehensive treatment approaches clinically, but we lack the human histologically proved data, whether DBBM bone substitute can be used safely when the tooth is exposed to OTM. Our main question is how orthodontic induced bone remodelling interferes with these graft particles, can they heal the same or even better compared to control sites. Tissue response might be different also in the case of the two test subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis with intrabony defect (Intrabony component ≥ 4mm, defect radiological angulation > 25°, 1 or max. 2 bony walls (no buccal bony wall), non-containing defect), no class III. furcation involved teeth
* Selected tooth must be in a traumatic occlusion or not in a gnathologically correct bite (migrated, elongated, tilted tooth, etc.).
* Patients must not be heavy smokers (<5 cigarettes/day).
* Full mouth plaque and bleeding scores (FMPS and FMBS) of <20% (O'Leary et al. 1972).
* The patient is able to comply with the study -related procedures (i.e. good level of oral hygiene, follow-up procedures).
* The patient is able to fully understand the nature of the study, signed informed consent.

Exclusion Criteria:

* Pregnant women.
* Participation in another clinical study within 30 days prior to study start.
* Alcoholism, drug dependency, heavy smoking (>5 cigarettes/day).
* Known infection with HIV, HBV, or HCV.
* Patients requiring chemo- or radiotherapy.
* Previous or current radiotherapy of the head.
* Uncontrolled or insulin-dependent diabetes mellitus
* Clinically relevant osteoporosis or systemic disease affecting bone metabolism
* Clinically relevant cardiovascular disease e.g., decompensated cardiac insufficiency, hemodynamically relevant heart valve defects, or myocardial infarction during the last three months.
* Clinically relevant blood coagulation disorder.
* Previous or current treatment with systemic corticosteroids (within 2 months prior to screening visit) of more than 5 mg/day prednisone equivalent.
* Previous or current therapy with bisphosphonates at least for 30 days within the last 12 months before screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Amount of newly formed bone by means of histomorphometry | 9 months postoperatively
  The percentage of newly formed bone of the former periodontal defect after a biopsy harvesting during a reentry surgery 9 months after the GTR intervention
Amount of graft material by means of histomorphometry | 9 months postoperatively
  The percentage of graft material (BioOss, Geistlich Pharma AG, Wolhusen) of the former periodontal defect after a biopsy harvesting during a reentry surgery 9 months after the GTR intervention
Amount of connective tissue by means of histomorphometry | 9 months postoperatively
  The percentage of connective tissue of the former periodontal defect after a biopsy harvesting during a reentry surgery 9 months after the GTR intervention

SECONDARY OUTCOMES:
CAL | 9 months postoperatively
  Clinical attachment level gain
PPD | 9 months postoperatively
  Pocket probing depth reduction
GR | 9 months postoperatively
  Change in gingival recession
Bone gain | 9 months postoperatively
  The absolute fill of the periodontal defect
Bone loss | 9 months postoperatively
  The change of the crestal bony wall
Intrabony fill | 9 months postoperatively
  The change of the intrabony component compared to the initial intrabony defect depth (in percentage)

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo MG, Carmagnola D, Berglundh T, Thilander B, Lindhe J. Orthodontic movement in bone defects augmented with Bio-Oss. An experimental study in dogs. J Clin Periodontol. 2001 Jan;28(1):73-80. doi: 10.1034/j.1600-051x.2001.280111.x. PMID 11142670
- [Background] Zucchelli G, De Sanctis M. A novel approach to minimizing gingival recession in the treatment of vertical bony defects. J Periodontol. 2008 Mar;79(3):567-74. doi: 10.1902/jop.2008.070315. PMID 18315442
- [Background] Reynolds MA, Aichelmann-Reidy ME, Branch-Mays GL, Gunsolley JC. The efficacy of bone replacement grafts in the treatment of periodontal osseous defects. A systematic review. Ann Periodontol. 2003 Dec;8(1):227-65. doi: 10.1902/annals.2003.8.1.227. PMID 14971256
- [Background] Reichert C, Deschner J, Kasaj A, Jager A. Guided tissue regeneration and orthodontics. A review of the literature. J Orofac Orthop. 2009 Jan;70(1):6-19. doi: 10.1007/s00056-009-0814-1. Epub 2009 Feb 5. English, German. PMID 19194672
- [Background] Cardaropoli D, Re S, Manuzzi W, Gaveglio L, Cardaropoli G. Bio-Oss collagen and orthodontic movement for the treatment of infrabony defects in the esthetic zone. Int J Periodontics Restorative Dent. 2006 Dec;26(6):553-9. PMID 17243328